CLINICAL TRIAL: NCT01863576
Title: Effects of Omega-3 Polyunsaturated Fatty Acid Supplementation on the Cytokine and Lipid Profiles in Patients With Chronic Chagas Cardiomyopathy: a Randomized Controlled Clinical Trial
Brief Title: Effects of Omega-3 Supplementation on the Cytokine and Lipid Profiles in Patients With Chronic Chagas Cardiomyopathy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Evandro Chagas Institute of Clinical Research (Other)
Collaborators: Andrea Silvestre de Sousa, MD PhD (Unknown); Alejandro Marcel Hasslocher, MD MSc PhD student (Unknown); Andrea Pereira de Souza, PhD (Unknown); Claudia Santos de Aguiar Cardoso, MSc (Unknown); Patricia Dias de Brito, PhD (Unknown); Pedro Emmanuel Alvarenga Americano do Brasil, MD PhD (Unknown); Roberta Olmo Pinheiro, PhD (Unknown); Roberto Magalhães Saraiva, MD PhD (Unknown); Sergio Salles Xavier, MD PhD (Unknown); Paula Simplicio da Silva, MSc PhD student (Unknown)
Responsible Party: Principal Investigator, Gilberto Marcelo Sperandio da Silva, PhD, Evandro Chagas Institute of Clinical Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 0037.0.009.000-10
Record Dates: First submitted 2013-05-22; First posted 2013-05-29 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Chagas Cardiomyopathy
Keywords: Chagas disease; Chagas Cardiomyopathy; Trypanosoma cruzi; Omega-3; Cytokines; Lipid profile; Nutritional assessment
MeSH Terms: conditions — Chagas Cardiomyopathy; Chagas Disease | interventions — Docosahexaenoic Acids; Fish Oils; Fatty Acids, Omega-3; Fatty Acids, Unsaturated; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 (Active Comparator): This group is receiving omega-3 supplement.
  Interventions: Dietary Supplement: Omega-3
- Oil Corn (Placebo Comparator): This group is receiving the placebo comparator.
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Omega-3 — The group omega-3 receives 5 capsules / day, each capsule containing 1100mg of lipids, and 600 mg of omega-3, 3g of omega-3 per day (1.8 g EPA and 1.2 g DHA) for a period of 8 weeks.
  Other Names: Oil fish; omega 3 fatty acids; polyunsaturated fatty acids
  Arms: Omega-3
Dietary Supplement: Placebo Comparator — The group placebo receives 5 capsules / day of corn oil containing 1100mg each, for a period of 8 weeks.
  Other Names: Oil Corn
  Arms: Oil Corn

SUMMARY:
The objective of this trial is to study the effects of omega-3 PUFA supplementation on the inflammatory response and lipid profile in patients with chronic Chagas cardiomyopathy.

Study Type: Interventional

Study Design: A total 40 patients will be randomly assigned into two parallel groups. The intervention will be treatment with omega-3 PUFAs at a dose of 3 g/day for 8 weeks, compared to placebo (corn oil). The primary endpoints will be the concentrations of inflammatory markers (IL-1, IL-2, IL-4, IL-6, IL-10, TNF-alpha, IFN-γ, and TGF-β). Secondary endpoints will be the fasting glucose, lipid, and anthropometric profiles.

DETAILED DESCRIPTION:
Several studies have shown the beneficial effects of polyunsaturated fatty acids on inflammatory processes, dyslipidemia, and cardiovascular diseases, there are no reports about food intake and PUFA supplementation in chronic Chagas cardiomyopathy patients. Thus, the objective of this study is to assess the effects of omega-3 PUFA supplementation on the lipid profile and the pro-inflammatory and anti-inflammatory cytokine profiles in chronic Chagas cardiomyopathy patients.

After patients are selected by cardiologists, they will be seen by study nutritionists, who will explain the study procedures to the patients and administer the free and informed consent form. The patients who agree to participate in the study will sign the consent form and undergo the initial assessment.

The following data will be collected and evaluated in the study: sociodemographic data (age, sex, ethnicity/race, education, and domicile), clinical data (functional class and vital signs), alcoholism, smoking, prescription drugs, 3-day food record, 24-hour recall, anthropometric assessment (height, weight, BMI, waist circumference, tricipital skinfold thickness, and arm circumference), lipid profile (total cholesterol, triglycerides, HDL-c, LDL-c, and VLDL-c), and cytokines (IL-1, IL-2, IL-4, IL-6, IL-10, TNF-alpha, IFN-γ, and TGF-β). Clinical, nutritional, and anthropometric assessments will take place immediately before starting the intervention and after 4 and 8 weeks during the study; lipid profile and cytokines will be evaluated before the intervention and at the end of 8 weeks. Each patient will be followed for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with Chagas Cardiomyopathy at stage B (no heart failure symptoms but with segmental or global left ventricular systolic dysfunction), stage C (symptomatic heart failure), or stage D (end-stage heart failure)), according to the current Brazilian Chagas' Disease Consensus;
* Subjects will include adults, men and women.

Exclusion Criteria:

* diarrheal disease;
* inflammatory bowel syndrome;
* diagnosis of diabetes or other endocrine pathologies;
* use of fibrates, niacin, or statins;
* use of anti-inflammatory drugs;
* pregnant and lactating women;
* vitamin mineral or omega-3 supplementation during the previous 30 days;
* hospital admission during the study;
* presence of cardiomyopathies other than Chagas Cardiomyopathy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cytokine profile | 8 weeks
  The primary endpoint of this study will be the cytokine profile. IL-1, IL-2, IL-4, IL-6, IL-10, TNF-alpha, IFN-γ, and TGF-β will be measured in the serum of patients using specific sandwich enzyme-linked immunosorbent assays. Capture and detection antibodies will be obtained from eBioscience (San Diego, CA, USA).

SECONDARY OUTCOMES:
Lipid profile | 8 weeks
  Total cholesterol, triglycerides, and high-density lipoprotein cholesterol (HDL-c) will be measured with enzymatic-colorimetric assays using Siemens reagents on a Siemens Dimension RXL chemistry analyzer (Siemens Healthcare Diagnostics, Tarrytown, NY, USA). Low-density lipoprotein cholesterol (LDL-c) and VLDL-c will be calculated according to the Friedewald equation

OTHER OUTCOMES:
Anthropometric measures | 8 weeks
  The anthropometric assessment will consist of body mass index (BMI), waist circumference, tricipital skinfold thickness, and arm circumference.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea S Sousa, MD PhD, Study Director — Evandro Chagas Institute of Clinical Research
Locations (1):
- Evandro Chagas Institute of Clinical Research, Rio de Janeiro, Br|rj, Brazil

REFERENCES:
- [Derived] Silva PSD, Mediano MFF, Silva GMSD, Brito PD, Cardoso CSA, Almeida CF, Sangenis LHC, Pinheiro RO, Hasslocher-Moreno AM, Brasil PEAAD, Sousa AS. Omega-3 supplementation on inflammatory markers in patients with chronic Chagas cardiomyopathy: a randomized clinical study. Nutr J. 2017 Jun 9;16(1):36. doi: 10.1186/s12937-017-0259-0. PMID 28599665
- [Derived] Silva PS, Sperandio da Silva GM, de Souza AP, Cardoso CS, Fonseca CA, Brito PD, Saraiva RM, Brasil PE, Pinheiro RO, Hasslocher-Moreno AM, Xavier SS, Sousa AS. Effects of omega-3 polyunsaturated fatty acid supplementation in patients with chronic chagasic cardiomyopathy: study protocol for a randomized controlled trial. Trials. 2013 Nov 11;14:379. doi: 10.1186/1745-6215-14-379. PMID 24216069